CLINICAL TRIAL: NCT05176522
Title: Motor REHAbilitation TEChnologies for CHIldren With Disability
Brief Title: Motor REHAbilitation TEChnologies for CHIldren With Disability: A Cross-European Survey
Acronym: RehaTech4Child
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Fondation Ildys (Other); BEaCHILD; France (Unknown); Salud de Madrid; Espagne (Unknown); National Clinic Center for Neuro-psychomotor Rehabilitation of Children (CNCRNC); Roumanie (Unknown); KU Leuven; Belgique (Unknown); Hôpital Nestlé CHUV; Suisse (Unknown)
Responsible Party: Sponsor
Other Study IDs: RehaTech4Child
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-06

CONDITIONS: Children With Disabilities; Motor Rehabilitation; Technologies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the RehaTech4Child survey led by EACD is to identify the digital technologies (e.g., robotic devices and treadmill systems, virtual reality and gaming systems, telehealth) that are used in clinical practices throughout Europe, and to know more about how rehabilitation professionals use or not use digital technologies in motor rehabilitation practices within the paediatric population. This knowledge would eventually help in designing the future technological developments based on the feedback from rehabilitation professionals.

ELIGIBILITY:
Inclusion Criteria:

* Rehabilitation professionals who use or not technologies in pediatric motor rehabilitation
* Practice in Europe

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Survey-takers across Europe who will participate in the online survey
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Access, frequency of use and intention to use of digital technologies by paediatric motor rehabilitation professionals A Cross-European Web survey | From Februray till June 2022
  To investigate the access to, the frequency of use and the intention to use digital technologies by paediatric motor rehabilitation professionals, and to assess their determinants

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ildys, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pons C, Brochard S, Grigoriu A, Newman CJ, Monbaliu E, Mensah-Gourmel J, Gaudin-Drouelle D, Toumi A, Konings M, de la Cruz J. Digital technologies for motor rehabilitation in children: protocol for a cross-sectional European survey. BMJ Open. 2023 Apr 25;13(4):e069034. doi: 10.1136/bmjopen-2022-069034. PMID 37185191